CLINICAL TRIAL: NCT04607200
Title: A Phase 2 Study Examining AGEN2034 as a Single-Agent and in Combination With AGEN1884 in Patients With Recurrent, Inoperable Angiosarcoma
Brief Title: AGEN2034 & AGEN1884 in Patients With Recurrent, Inoperable Angiosarcoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Strategic business decision
Sponsor: Agenus Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C-550-02
Record Dates: First submitted 2020-10-16; First posted 2020-10-29 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Angiosarcoma
MeSH Terms: conditions — Hemangiosarcoma | interventions — balstilimab; spartalizumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Monotherapy (Experimental): AGEN2034 - dose of 3 mg/kg IV every 2 weeks for up to 24 months
  Interventions: Drug: AGEN2034
- Combination Therapy (Experimental): AGEN2034 - dose of 3 mg/kg IV every 2 weeks + AGEN1884 - dose of 1 mg/kg IV every 6 weeks (following AGEN2034 infusion), for up to 24 months
  Interventions: Drug: AGEN2034; Drug: AGEN1884

INTERVENTIONS:
Drug: AGEN2034 — Anti-PD-1 Monoclonal Antibody
  Other Names: Anti-PD-1
Drug: AGEN1884 — Anti-CTLA-4 Monoclonal Antibody
  Other Names: Anti-CTLA-4
  Arms: Combination Therapy

SUMMARY:
This Phase 2, open-label study is designed to examine the efficacy and safety of single-agent AGEN2034 and combination AGEN2034 + AGEN1884 in patients with recurrent, inoperable or metastatic Angiosarcoma (AS).

DETAILED DESCRIPTION:
This Phase 2, open-label study is designed to examine the efficacy and safety of single-agent AGEN2034 and combination AGEN2034 + AGEN1884 in patients with recurrent, inoperable or metastatic AS.

Three cohorts will be enrolled into 2 Parts of the study as follows:

Part 1

* Cohort 1: Qualifying patients that are checkpoint inhibitor naïve will be enrolled into single-agent AGEN2034
* Cohort 2: Qualifying patients that are inhibitor (PD-1/L1) resistant will be enrolled into combination AGEN2034 + AGEN1884

Part 2

• Cohort 3: Qualifying patients that are checkpoint inhibitor naïve will be enrolled into combination AGEN2034 + AGEN1884. Part 2 will begin enrollment after enrollment in Part 1 is completed

The study will be conducted in 2 parts:

In Part 1, checkpoint inhibitor naïve patients will be treated with single-agent AGEN2034 (Cohort 1) and patients resistant to PD-1/PD-L1 (defined as prior progression on PD 1/PD-L1 treatment) will be treated with combination of AGEN2034+AGEN1884 (Cohort 2). Patients from Cohort 1 who experience PD may be considered (as PD-1 resistant) for transition to Cohort 2.

In Part 2, the study will enroll checkpoint inhibitor naïve patients for treatment with combination AGEN2034+AGEN1884 (Cohort 3). Part 2 will begin enrollment after enrollment in Part 1 is completed.

All patients will receive study treatment for up to 2 years until confirmed disease progression, unacceptable toxicity, or until the patient wishes to withdraw consent for any reason. Patients will be followed for safety at 30 and 90 days, and for survival every 2 months for at least 12 months from their last dose of study treatment. Each treatment cycle will be 6 weeks.

An IRC will be established to adjudicate tumor response based on imaging studies, photography, and clinical response. The primary endpoints will be based on the IRC assessment of response per RECIST v1.1.

ELIGIBILITY:
Inclusion Criteria

To be eligible for this study, patients must meet the following inclusion criteria:

1. Histologically confirmed AS not amenable to curative intent surgery
2. Prior treatment history for AS

   1. Cohort 1 and Cohort 3

      * Patients who previously received and progressed after at least 1 prior therapy for AS.
      * Checkpoint inhibitor (PD-1/PD-L1/CTLA-4) naïve
   2. Cohort 2

      * Patients who previously received and progressed on or after at least 1 prior therapy for AS
      * Prior treatment must include PD-1 or PD-L1 inhibitor such as nivolumab, pembrolizumab, atezolizumab, durvalumab, AGEN2034, or other, given either as the most recent treatment or earlier. Note: Confirmation of PD is required after treatment with prior checkpoint inhibitors
      * CTLA-4 inhibitor naïve
3. ≥ 18 years of age.
4. At least one lesion measurable, either radiologically (computed tomography [CT], magnetic resonance imaging [MRI]) and/or using color photography with a ruler, as per RECIST v1.1
5. Have a life expectancy of ≥ 3 months and an Eastern Cooperative Oncology Group Performance Status of 0 to 1
6. Resolution of all acute AEs resulting from prior cancer therapies to National Cancer Institute Common Terminology Criteria for Adverse Events Version 5.0 Grade ≤ 1
7. Have adequate organ function as indicated by the following laboratory values:

   1. Adequate hematological function defined by absolute neutrophil count > 1.5 × 10^9/L, platelet count > 75 × 10^9/L, and hemoglobin > 8 g/dL (without transfusions, within

      1 week of first dose)
   2. Adequate hepatic function based by a total bilirubin level ≤ × 1.5 the upper limit of normal (ULN), aspartate aminotransferase level ≤ 2.5 × ULN, alanine aminotransferase level ≤ 2.5 × ULN, alkaline phosphatase ≤ 2.5 × ULN, and albumin

      ≥ 3.0 mg/dL
   3. Adequate renal function defined as creatinine ≤ 1.5 × ULN OR measured or calculated creatinine clearance ≥ 40 mL/minute per Institutional standard. Assessment methods should be recorded
   4. Adequate coagulation defined by international normalized ratio or prothrombin time ≤ 1.5 × ULN (unless the patient is receiving anticoagulant therapy); and activated partial thromboplastin time ≤ 1.5 × ULN (unless the patient is receiving anticoagulant therapy)
8. Willing to undergo mandatory fresh tumor biopsy, from a site not previously irradiated (unless progressed after radiation treatment) Note: Tissue from core, or punch excisional biopsy, or from resection is required
9. Women of child-bearing potential (WCBP) must have a negative serum pregnancy test at Screening (within 72 hours prior to first dose of study medication)

   Note: Non-childbearing potential is defined as 1 of the following:
   1. ≥ 45 years of age and has not had menses for > 1 year
   2. Amenorrheic for > 2 years without a hysterectomy and/or oophorectomy and follicle-stimulating hormone value in the postmenopausal range upon pre-study (Screening) evaluation
   3. Status is post hysterectomy, oophorectomy, or tubal ligation
10. WCBP must be willing to use highly effective contraception throughout the study, starting with the Screening Visit through 90 days after the last dose of study treatment
11. Male patients with a female partner(s) of childbearing potential must agree to use highly effective contraceptive measures throughout the study starting with the Screening Visit through 90 days after the last dose of study treatment is received. Males with pregnant partners must agree to use a condom; no additional method of contraception is required for the pregnant partner Note: Abstinence is acceptable if this is the established and preferred contraception method for the patient
12. Willingness and ability to consent to participate in study and comply with all study procedures

Exclusion Criteria

To be eligible for this study, patients must not have any of the following exclusion criteria:

1. Is currently participating and receiving study therapy or has participated in a different study of an investigational agent and received study therapy or used an investigation device within 3 weeks of the first dose of treatment
2. Has an inadequate washout period prior to first dose of study drug defined as:

   1. < 3 weeks from last dose of prior systemic cytotoxic chemotherapy or biological therapy
   2. < 3 weeks from last radiation therapy
   3. < 4 weeks from major surgery
3. Known severe (Grade ≥ 3) hypersensitivity reactions to fully human mAbs, antibody, or severe reaction to immuno-oncology agents, such as colitis or pneumonitis requiring treatment with steroids
4. Has received systemic corticosteroid therapy ≤ 7 days prior to the first dose of study treatment or receiving any other form of systemic immunosuppressive medication (corticosteroid use on study for management of immune-related AEs, and/or a premedication for intravenous (IV) contrast allergies/reactions is allowed). Patients who are receiving daily corticosteroid replacement therapy are an exception to this rule. Daily prednisone at doses of up to 7.5 mg or equivalent hydrocortisone dose are examples of permitted replacement therapy
5. Known central nervous system tumor, metastasis(es), and/or carcinomatous meningitis identified either on the Baseline brain imaging obtained during the Screening Period or identified prior to consent Note: Patients with history of brain metastases that have been treated may participate provided they show evidence of stable supra-tentorial lesions at Screening (based on 2 sets of brain images, performed ≥ 4 weeks apart, and obtained after the brain metastases treatment).

   In addition, any neurologic symptoms that developed either as a result of the brain metastases or their treatment must have resolved or be minimal and be expected as sequelae from treated lesions. For individuals who received steroids as part of brain metastases treatment, high-dose steroids must be discontinued ≥ 7 days prior to first dose of study drug but may be continued if ≤ 5 mg/day (prednisone)
6. Has active or history of autoimmune disease requiring immunosuppressive systemic treatment (e.g. modifying agents, corticosteroids or immunosuppressive drugs) within previous 2 years Note: Thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency is not considered a form of immunosuppressive systemic treatment.

   Note: Patients with Type 1 diabetes, vitiligo, psoriasis, hypo-, or hyperthyroid disease not requiring immunosuppressive treatment are eligible
7. Has had an allogeneic tissue/solid organ transplant
8. Has or had interstitial lung disease or has had a history of pneumonitis anaphylaxis, or uncontrolled asthma that has required oral or IV corticosteroids
9. Active infection requiring IV systemic therapy
10. Known history of HIV type 1 or 2 antibodies
11. Known active infection with hepatitis B and/or hepatitis C virus
12. History of seizure disorders
13. Clinically significant cardiovascular disease: cerebral vascular accident/stroke or myocardial infarction within 6 months of enrollment, unstable angina, congestive heart failure (New York Heart Association class ≥ II), or serious uncontrolled cardiac arrhythmia requiring medication
14. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate, in the opinion of the treating Investigator
15. Psychiatric or substance abuse disorder that would interfere with cooperation with the requirements of the study
16. Legally incapacitated or has limited legal capacity
17. Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-02 (Estimated); Primary Completion 2021-09-13 (Actual); Study Completion 2021-09-13 (Actual)

PRIMARY OUTCOMES:
Response rate of single-agent AGEN2034 and combination AGEN2034 + AGEN1884 | 48 months
  To evaluate the response rate of single-agent AGEN2034 and combination AGEN2034 + AGEN1884 per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) in patients with recurrent angiosarcoma

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Agenus Inc.